CLINICAL TRIAL: NCT04583202
Title: Evaluation of the Nasal and Conjunctival Response in Subjects Allergic to Birch Pollen in the ALYATEC Environmental Exposure Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: ALY-004
Record Dates: First submitted 2020-09-30; First posted 2020-10-12 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2020-11

CONDITIONS: Allergic Rhinitis; Allergy to Pollen; Rhinoconjunctivitis
Keywords: Environmental Exposure Chamber; Allergen Exposure Chamber; Allergen provocation test; Birch pollen
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo exposure (Placebo Comparator): All patients undergo 2 placebo exposures
  Interventions: Other: Exposure to placebo
- Birch Pollen Exposure (Experimental): All patients undergo 4 allergen exposures
  Interventions: Other: Exposure to allergen

INTERVENTIONS:
Other: Exposure to placebo — Patients are exposed to a placebo for 4h in the Alyatec EEC
  Arms: Placebo exposure
Other: Exposure to allergen — Patients are exposed to birch pollen allergens for 4h in the Alyatec EEC
  Arms: Birch Pollen Exposure

SUMMARY:
The aim of this study is to assess the nasal and conjunctival response in subjects allergic to birch pollen during controlled exposures in the ALYATEC environmental exposure chamber (EEC)

DETAILED DESCRIPTION:
This is a single-center, single-blind, placebo-controlled study. The first part of the study consists of 6 exposure sessions in Alyatec EEC, including placebo and birch pollen allergen exposures.

The second part of the study involves in-field evaluations of rhinitis and conjunctivitis symptoms during birch pollen season.

Alyatec environmental exposure chamber, also called allergen challenge chamber, allows to evaluate allergic symptoms in standardized and reproducible conditions. All the metrological parameters (temperature, air flow, hygrometry ...) are controlled as well as the allergen concentration diffused in the room.

This enables to induce and observe rhinitis, conjunctivitis and asthma symptoms for up to 20 patients at the same time, in a reproducible way and without the potential perturbations or contaminations of the natural environment.

The current study aims to get specific information about allergic symptoms induced in the Alyatec EEC chamber in patients sensitized to birch pollen allergen.

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of allergic rhinitis to birch pollen for at least 2 consecutive pollen seasons requiring the taking of a symptomatic drug with or without associated asthma
* Positive skin prick tests for birch pollen (> 3 mm)
* IgE specific to birch > 0.75 kUI / L.
* Positive unit rapid nasal provocation test for birch pollen
* Subjects having signed informed consent
* Subjects affiliated to a social security scheme
* Subjects able to understand and complete the procedures related to the study
* Women of childbearing potential should have a negative pregnancy test throughout the study period with effective contraception

Exclusion Criteria:

* Specific immunotherapy (SIT) for birch allergens for more than a month in the 3 years preceding the screening
* Current use of Specific immunotherapy for another allergen
* Medical history of anaphylaxis following exposure to birch pollen
* Medical history of anaphylaxis linked to another allergen in the last 6 weeks
* Nasal polyps, nasal septum deviation or diagnosis of non-allergic rhinitis
* Subjects allergic to indoor environmental allergens (cat allergens, mold, dust mites) with - Obvious exposure to these allergens.
* Uncontrolled allergic pathology (rhinitis, conjunctivitis)
* Forced expiratory volume in 1 second (FEV1) <70% of predicted normal values
* Moderate to severe asthma (GINA 3 to 5)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | 4 hours exposure
  To assess the nasal response during exposure to birch allergens compared to placebo in the ALYATEC EEC.

SECONDARY OUTCOMES:
Visual Analogue Scale for rhinitis | 4 hours exposure
  To evaluate the intensity of the nasal response during exposure to birch allergens compared to placebo in the ALYATEC EEC.
Total Nasal Symptom Score | 4 hours exposure
  To evaluate the intensity of the nasal response during exposure to birch allergens compared to placebo in the ALYATEC EEC.
Visual Analogue Scale for conjunctivitis | 4 hours exposure
  To evaluate the intensity of the conjunctival response during exposure to birch allergens compared to placebo in the ALYATEC EEC.
Total Ocular Symptom Score | 4 hours exposure
  To evaluate the intensity of the conjunctival response during exposure to birch allergens compared to placebo in the ALYATEC EEC.
Peak Nasal Inspiratory Flow | 4 hours exposure
  To evaluate the nasal obstruction during exposure to birch allergens compared to placebo in the ALYATEC EEC.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr., Principal Investigator — Alyatec
Locations (1):
- Alyatec, Strasbourg, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alyatec website — https://www.alyatec.com/en/